CLINICAL TRIAL: NCT02419144
Title: Good Oral Health - A Bi-level Intervention to Improve Older Adult Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Susan Reisine, Professor Emeritus, UConn Health
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 14-188-6
Record Dates: First submitted 2015-04-08; First posted 2015-04-17 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Gingivitis
Keywords: older adults;; oral hygiene;; adapted motivational interviewing
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMI followed by campaigns (Active Comparator): Behavioral interventions
  Interventions: Behavioral: AMI and campaigns
- Campaigns followed by AMI (Active Comparator): Behavioral interventions
  Interventions: Behavioral: AMI and campaigns

INTERVENTIONS:
Behavioral: AMI and campaigns — The intervention we are proposing is a tailored bi-level intervention with two components, an individual level component (component A) with tailored messages based on performance on clinical assessment results, ADLs and cognitive domains in the survey delivered through adapted motivational interviewing with practice to mastery (AMI-PM); , and a building level campaign (component B) for those enrolled in the study (but open to all building residents that includes building tailored messages based on cognitive domains and skills reinforcement through Practice to Mastery.

SUMMARY:
This study will test an intervention designed to change oral health norms and reduce disparities in oral health among vulnerable adults residing in publicly funded senior housing in Central Connecticut. The intervention model is based on Fishbein modified theory of reasoned action operationalized through Adapted Motivational Interviewing and Practice to Mastery. The intervention includes two components: 1) a face to face administration of the Adapted Motivational Interviewing and Practice to Mastery, a participatory counseling model, and 2) a targeted building level campaign consisting of three half-day oral health events with skills development through practice to mastery to parallel the individual intervention, all based on the study's conceptual model. The study uses a modified fractional factorial design to evaluate the face to face and campaign components separately and in different additive sequences. Six buildings will be paired in three dyads. The buildings in each dyad will be randomized to either having the Adapted Motivational Interviewing and Practice to Mastery intervention first followed by campaigns or to having the campaigns first followed by Adapted Motivational Interviewing and Practice to Mastery. Seventy-five residents will be recruited in each building for a total of 450 participants. There will be four assessments:

1. T0 will include a survey, oral hygiene skills assessment and clinical assessment of the Gingival Index and Plaque Score. The survey will provide data on the conceptual domains that are the target of the tailored intervention
2. T1 will follow the AMI-PM or CA+PM (depending on condition) and will include the survey, oral hygiene skills assessment and clinical assessment of the Gingival Index and Plaque Score. This assessment will occur 1-2 months after the initial intervention
3. T2 will follow the AMI-PM or CA+PM and will include the survey, oral hygiene skills assessment and clinical assessment of the Gingival Index and Plaque Score. This assessment will occur 6 months after the initial intervention
4. T3 will include oral hygiene skills assessment and clinical assessment of the Gingival Index and Plaque Score. This will occur 15-18 months after study entry. We will use general linear mixed models (GLMM) or general estimating equations (GEE), respectively, to fit a model with intervention and period effects using the MIXED procedure in SAS.

ELIGIBILITY:
Inclusion Criteria:

1. Disabled children and adults aged 18 years and above, and adults 62 and above, including both male and female building residents, and minorities and non-minorities;
2. Permanent residence in sample buildings;
3. Independent of conservator;
4. Must be able to speak English or Spanish;
5. Judged competent to participate (based on ability to respond correctly to key questions about information covered during administration of informed consent.
6. Have two or more remaining natural teeth.

Exclusion Criteria:

1. Considered by research staff to be cognitively unable to give informed consent;
2. Exhibition of continued disruptive behavior while participating in the project;
3. History of infective endocarditis, prosthetic cardiac valve replacement, insertion of an arterial stent in past 6 months, myocardial infarction (heart attack) in past 6 months
4. under conservatorship
5. fewer than two natural teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Plaque scores from preintervention, at one month post intervention, 3 months post intervention and 6 months | pre-intervention, one month, 3 month and 6 month follow-up
  We will use a plaque scoring scheme developed by O'Leary (O'Leary, Drake, Naylor, 1972). This index consists of dichotomous presence or absence scores for plaque on each tooth surface. The supragingival bacterial plaque will be assessed with the use of erythrosine disclosing solution in six surfaces of each tooth. The non-toxic vegetable-based solution will be applied to the teeth by the examining hygienist. The number of surfaces stained red will be calculated over the total number of surfaces and the plaque score will be expressed as a percentage of surfaces with plaque as a ratio. We used this measure in the pilot study and demonstrated significant reductions in plaque after the intervention.
Change in Gingival Index from preintervention, at one month post intervention, 3 months post intervention and 6 months | pre-intervention, one month, 3 month and 6 month follow-up
  The Gingival Index (GI) (Loe & Silness, 1963) will be used to assess the gingival status related to six surfaces of each tooth. Each surface is scored for gingival inflammation: 0=no visual signs of inflammation; 1=slight change in color and texture of the gingiva but no bleeding; 2=visual sign of inflammation and bleeding upon swiping; 3=overt inflammation and spontaneous bleeding. The index is calculated by summing each surface GI and dividing by the total number of surfaces (mean value). Individual scores are summed to obtain a mean.

SECONDARY OUTCOMES:
Change in Oral Health Related Quality of Life Change from preintervention, at one month post intervention, 3 months post intervention and 6 months | pre-intervention, one month, 3 month and 6 month follow-up
  ): We will use the General (Geriatric) Oral Health Assessment Inventory (GOHAI), a commonly used 12-item measure initially developed for older adults that has been used with low income populations (Atchison & Dolan, 1990).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Reisine, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Reisine S, Schensul JJ, Salvi A, Grady J, Ha T, Li J. Oral health-related quality of life outcomes in a randomized clinical trial to assess a community-based oral hygiene intervention among adults living in low-income senior housing. Health Qual Life Outcomes. 2021 Sep 28;19(1):227. doi: 10.1186/s12955-021-01859-w. PMID 34583694
- [Derived] Schensul J, Reisine S, Salvi A, Ha T, Grady J, Li J. Evaluating mechanisms of change in an oral hygiene improvement trial with older adults. BMC Oral Health. 2021 Jul 21;21(1):362. doi: 10.1186/s12903-021-01701-1. PMID 34289839
- [Derived] Reisine S, Schensul JJ, Salvi A, Grady J, Ha T, Li J. Does sequencing matter? A cross-over randomized trial to evaluate a bi-level community-based intervention to improve oral hygiene among vulnerable adults. Community Dent Oral Epidemiol. 2022 Aug;50(4):270-279. doi: 10.1111/cdoe.12663. Epub 2021 Jun 6. PMID 34091935
- [Derived] Schensul JJ, Salvi A, Ha T, Grady J, Li J, Reisine S. Evaluating Cognitive/Emotional and Behavioral Mediators of Oral Health Outcomes in Vulnerable Older Adults. J Appl Gerontol. 2022 Jan;41(1):187-197. doi: 10.1177/0733464820974920. Epub 2020 Dec 8. PMID 33292050
- [Derived] Schensul J, Reisine S, Grady J, Li J. Improving Oral Health in Older Adults and People With Disabilities: Protocol for a Community-Based Clinical Trial (Good Oral Health). JMIR Res Protoc. 2019 Dec 18;8(12):e14555. doi: 10.2196/14555. PMID 31850853

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT02419144/Prot_SAP_ICF_000.pdf